CLINICAL TRIAL: NCT01130259
Title: An Open-Label, Expanded Access Protocol of Iniparib in Combination With Gemcitabine/Carboplatin in Patients With ER-, PR-, and HER2-Negative Metastatic Breast Cancer
Brief Title: An Open-Label, Expanded Access Protocol of Iniparib Breast Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: EFC11614; 2010EAP (Other: BiPar)
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: mTNBC; triple negative breast cancer; metastatic triple negative breast cancer; metastatic breast cancer that is ER-, PR-, and HER2-negative
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — iniparib

INTERVENTIONS:
Drug: iniparib — 5.6 mg/kg as a 60 (±10) minutes IV infusion. Administered on Days 1, 4, 8, and 11 of each 21 day cycle.
  Other Names: BSI-201

SUMMARY:
The following trial is designed to offer pre-approval drug access to iniparib in combination with gemcitabine and carboplatin in order to provide potential clinical benefit to patients with ER-, PR-, and HER2-negative metastatic breast cancer. This follows an ongoing Phase 3, multi-center, open-label, randomized study of gemcitabine/carboplatin, with or without iniparib, in patients with ER-, PR-, and HER2-negative metastatic breast cancer (protocol 20090301).

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented breast cancer (either primary or metastatic site) that is ER-negative, PR-negative, and HER2 non-over expressing by immunohistochemistry (0, 1) or in situ hybridization (ISH) including; fluorescence (FISH) in situ hybridization / chromogenic in situ hybridization (CISH) with a ratio < 2.0
* One to three prior chemotherapy regimens in the metastatic setting. Prior adjuvant/neoadjuvant therapy is allowed. Prior Gemcitabine and/or Platinum agents are allowed.
* Metastatic breast cancer (Stage IV)
* Female, ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Organ and marrow function as follows: absolute neutrophil count (ANC) ≥1500/mm3, platelets ≥100,000/dL, hemoglobin ≥9 g/dL, bilirubin ≤1.5 mg/dL, serum creatinine ≤1.5 mg/dL or creatinine clearance ≥60 mL/min, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal if no liver involvement or ≤5 times the upper limit of normal with liver involvement
* For women of child bearing potential, documented negative pregnancy test within two weeks of EAP entry and agreement to acceptable birth control during the duration of the EAP therapy
* Capability to understand and comply with the protocol and signed informed consent document

Exclusion Criteria:

* Systemic anticancer therapy within 14 days of the first dose of study drug
* Has not recovered to grade ≤1 from adverse events (AEs) per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v3.0, with the exception of alopecia, related to anticancer therapy prior to the first dose of study drug
* Major medical conditions that might affect EAP participation (e.g. uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection, cardiac disease)
* Brain metastases requiring steroids or expected to require other therapeutic intervention during study participation, including WBRT and intrathecal therapy. Patients must be > 21-days from neurosurgical intervention
* Pregnant or breastfeeding
* Inability or unwillingness to abide by the EAP protocol or cooperate fully with the investigator or designee

Enrollment is limited and will be determined by a validated Random-Selection Process administered by NORD (National Organization of Rare Disorders).

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi